CLINICAL TRIAL: NCT01306318
Title: A Clinical Study in Healthy Male Volunteers to Compare the Bioequivalence of Fixed Dose Combination of Eperisone Hydrochloride 50mg Plus Diclofenac Sodium 50mg as Capsule With Eperisone Hydrochloride 50mg and Diclofenac Sodium 50mg Tablets Under Fasting Conditions
Brief Title: A Clinical Study in Healthy Male Volunteers to Compare the Bioequivalence of Fixed Dose Combination of Eperisone Hydrochloride 50mg Plus Diclofenac Sodium 50mg as Capsule With Eperisone Hydrochloride 50mg and Diclofenac Sodium 50mg Tablets Under Fasting Conditions (Study 013-10)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eisai Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 013-10
Record Dates: First submitted 2011-02-24; First posted 2011-03-01 (Estimated); Last update posted 2015-11-17 (Estimated); Status verified 2015-11

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — eperisone; Diclofenac

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: eperisone hydrochloride plus diclofenac sodium capsule
- 2 (Active Comparator)
  Interventions: Drug: eperisone hydrochloride tablet and diclofenac sodium tablet

INTERVENTIONS:
Drug: eperisone hydrochloride plus diclofenac sodium capsule — Single dose of fixed dose capsule formulation of eperisone hydrochloride 50 mg plus diclofenac sodium 50 mg to be given in healthy volunteers in fasting conditions
  Arms: 1
Drug: eperisone hydrochloride tablet and diclofenac sodium tablet — Single dose of eperisone hydrochloride 50 mg as tablet formulation and diclofenac sodium 50 mg as tablet formulation to be given in healthy volunteers in fasting conditions
  Arms: 2

SUMMARY:
The primary objective of this study is to compare the bioavailabilities of a single fixed dose combination of eperisone 50 mg plus diclofenac 50 mg capsules with the bioavailabilities of eperisone 50 mg tablets and diclofenac 50 mg tablets in healthy human adult male subjects under fasting conditions.

DETAILED DESCRIPTION:
The primary objective of this study is to compare the single-dose oral bioavailabilities of eperisone and diclofenac from Epry-D (containing eperisone hydrochloride 50 mg and diclofenac sodium 50 mg) capsules of Eisai Pharmaceuticals India Private Limited, India with those from Epry (eperisone hydrochloride) 50 mg tablets of Eisai Pharmaceuticals India Pvt. Ltd., and voltaren (diclofenac sodium) 50 mg tablets of Novartis Pharmaceuticals Ltd., India in healthy human adult male subjects under fasting conditions. The secondary objective of this study is to monitor the safety and tolerability of a single dose of eperisone hydrochloride 50 mg and diclofenac sodium 50 mg formulation when administered in healthy human adult male subjects under fasting conditions. The participants will be screened for demographic data, medical history, general physical examination, 12-lead electrocardiogram (ECG), chest X-ray (Posterior to Anterior view), hematology, clinical bio- chemistry, serology, urine analysis, tests for alcohol and drugs of abuse. A total of 24 healthy adult male volunteer participants will be housed in the clinical study facility at least 11 hours before administration of the Investigational Product (IP) and will continue to remain in the clinical study facility for at least 12 hours after administration of the IP in each study period. After overnight fasting for at least 10 hours, either one Epry-D capsule or one Epry 50 mg tablet and one Voltaren 50 mg tablet will be administered orally to each participant in sitting posture, with 240 plus or minus 2 mL of water at room temperature, in each study period, as per the randomization schedule. Administration of the IP will be performed by trained study personnel. Dosing activity will be followed by mouth check to assess the compliance to dosing. A total of 22 (6 mL) blood samples will be collected from each subject in pre-specified vacuum tubes containing K2 EDTA in each study period.

ELIGIBILITY:
Inclusion Criteria

* Normal healthy human adult male volunteers between 18-45 years (both ages inclusive) of age, who have given written informed consent and are willing to participate in the study.
* Volunteer having Body Mass Index of 18.50 to 24.90 Kg/m2 (both inclusive).
* Volunteer with no evidence of underlying disease during the pre-study screening, medical history, physical examination and laboratory investigations performed within 21 days prior to commencement of the study
* Volunteer whose pre-study screening laboratory tests are either normal or within acceptable limits or are considered by the Investigator to be of no clinical significance with respect to his participation in the study.
* Volunteer with negative test for alcohol and drugs of abuse, hepatitis B and C and who is negative or nonreactive for antibodies to human immunodeficiency virus (HIV) 1 and 2 and rapid plasma reagin (RPR).
* Volunteer having a 12 lead electrocardiogram (ECG) recording within normal limits.
* Volunteer with normal chest X-ray taken within 6 months before the day of dosing.
* Volunteer will be available for the entire study period and is capable of understanding and communicating with the investigators and clinical study facility staff.

Exclusion Criteria

* Volunteer who is allergic to eperisone and/or diclofenac or any component of the formulation and to any other related drug.
* Volunteer with history or presence of significant cardiovascular, respiratory, hepatic, renal, hematological, gastrointestinal, endocrine, immunologic, dermatologic, neurological or psychiatric disease.
* More specifically, volunteer with history or presence of the following significant conditions:

  1. Alcohol dependence, alcohol abuse or drug abuse within the past one year, recent or current alcohol abuse (> 5 units/week, 1 unit= 10 mL or 8 g of pure alcohol) or suspected abuse.
  2. History of chronic smoking (more than 10 units per day of cigarettes, bidis, or any other form) or chronic consumption of tobacco products.
  3. Asthma, urticaria or other allergic type reactions after taking any medication.
  4. Clinically significant illness within 4 weeks before the start of the study.
  5. Hypersensitivity to heparin.
* History of clinically relevant allergy (except for untreated, asymptomatic, seasonal allergies at time of dosing) or any allergic reactions to any drugs.
* History of Vascular collapse.
* Volunteer who is scheduled for surgery within 7 days after study completion.
* Volunteer who, through completion of any other clinical or bioequivalence study or otherwise would have donated in excess of 350 mL of blood in the last 90 days.
* Volunteer who has taken prescription medication or over-the-counter products (including vitamins and products from natural origin) within 14 days prior to administration of IP in period 1, including topical medication meant for systemic absorption.
* Volunteer who was hospitalized within 28 days prior to administration of the study medication.
* Volunteer with pulse rate less than 60/min or more than 100/min.
* Volunteer with history of difficulty in swallowing.
* Volunteer who has unsuitable veins for repeated venipuncture.
* Any abnormal laboratory value or physical finding which may interfere with the interpretation of test results or cause a health hazard for the volunteer if he participates in the study.

Volunteer who has

* Systolic blood pressure less than 90 mm of Hg or more than 150 mm of Hg
* Diastolic blood pressure less than 60 mm of Hg or more than 90 mm of Hg. Minor deviations (2-4 mm of Hg) at check-in may be acceptable at the discretion of the Investigator.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2011-02; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Oral bioavailabilities: Maximum Concentration (Cmax) of eperisone and diclofenac fixed dose capsules versus eperisone & diclofenac tablets | 12 hours post dose
  Compare single-dose oral bioavailabilities (Cmax) of eperisone and diclofenac fixed dose capsules with eperisone & diclofenac tablets. Cmax is defined as the maximum observed concentration in plasma.

SECONDARY OUTCOMES:
Safety & tolerability (total number of subjects reporting adverse events) of single dose of fixed dose combination of eperisone and diclofenac in fasting conditions | 10 days
  Safety & tolerability measured as total number of participants reporting adverse events of single doses and fixed dose combination of eperisone and diclofenac in fasting conditions.

CONTACTS AND LOCATIONS:
Overall Officials: Suyog Mehta, Study Director — General Manager Medical & Regulatory Affairs, Eisai Pharmaceuticals India Private Limited, Mumbai, MS, India
Locations (1):
- Manipal AcuNova KH Clinical Research Center, Manipal, Karnataka, India